CLINICAL TRIAL: NCT03638479
Title: Utilizing Smart Devices to Identify New Phenotypical Characteristics in Movement Disorders
Status: Completed | Type: Observational
Sponsor: Universität Münster (Other)
Responsible Party: Principal Investigator, Julian Varghese, Principal Investigator, Universität Münster
Other Study IDs: VA111809
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Essential Tremor; Movement Disorders; Parkinson's Syndrome; Atypical Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's Disease: Participant's diagnosed with Parkinson's Disease
  Interventions: Other: Data Capture
- Essential Tremor: Participant's diagnosed with Essential Tremor or other Movement Disorders
  Interventions: Other: Data Capture
- No Parkinson's Disease and No Essential Tremor: Participant's with no diagnosis of PD, ET or other Movement Disorders
  Interventions: Other: Data Capture

INTERVENTIONS:
Other: Data Capture — This is no intervention. Participants of all groups will receive data Capture with smartphones, smartwatches and tablets.

SUMMARY:
This observational and experimental study seeks to establish a Smart Device System (SDS) to monitor high-resolution handtremor-based data using Smartphones, SmartWatches and Tablets. By doing this, movement data will be analyzed in depth with advanced statistical and Deep-Learning algorithms to identify new clinical phenotypical characteristics Parkinson's Disease and Essential Tremor.

DETAILED DESCRIPTION:
Current smart devices as smartphones and smartwatches have reached a level of technical sophistication that enables high-resolution monitoring of movements not only for everyday sports activities but also for movement disorders. Tremor-related diseases as Parkinson's Disease (PD) and Essential Tremor (ET) are two of the most common movement disorders. Disease classification is primarily based on clinical criteria and remains challenging. The primary goal of this study is to identify new phenotypical characteristics based on the captured movement data by the tremor-capturing smartwatches and tablets and smartphone-based questionnaires.

The system will be applied and analyzed within an experimental and observational setting and only captures from patients, which have received informed consent. Within the study period, the SDS is not intended as clinical diagnostic support for physicians and will be not be used as medical device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's Disease (ICD-10-GM G20.-) or Essential Tremor (G25.0)
* Comparison group: Other movement disorders including atypical Parkinsonian disorders and healthy participants

Exclusion Criteria:

* Unable to obtain informed consent
* Skin-related conditions at one of the wrists or any other medical conditions that could harm the participant's health by wearing the smartwatch at both wrists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who attend the ambulatory clinicic for movement disorders at the University Hospital Münster will be asked for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acceleration data in all three axes (x,y,z) measured at both wrists via Smartwatches during 10 minutes of neurological examination. Aggregated data: Mean Frequency and Amplitude of Tremor. | 2018-2020
  The raw time series data (acceleration data) and the aggregated data will be analyzed to train a neural network to classify the participant's movement disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Varghese, MD, Principal Investigator — WWU Münster, Institut für Medizinische Informatik
Locations (1):
- Institute of Medical Informatics, University of Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Purk M, Fujarski M, Becker M, Warnecke T, Varghese J. Utilizing a tablet-based artificial intelligence system to assess movement disorders in a prospective study. Sci Rep. 2023 Jun 26;13(1):10362. doi: 10.1038/s41598-023-37388-3. PMID 37365210
- [Derived] Varghese J, Niewohner S, Soto-Rey I, Schipmann-Miletic S, Warneke N, Warnecke T, Dugas M. A Smart Device System to Identify New Phenotypical Characteristics in Movement Disorders. Front Neurol. 2019 Jan 30;10:48. doi: 10.3389/fneur.2019.00048. eCollection 2019. PMID 30761078